CLINICAL TRIAL: NCT00613106
Title: Double-Blind Follow-On Safety Study of HZT-501 (Ibuprofen 800 mg/Famotidine 26.6 mg)in Subjects Who Have Completed Participation in Horizon Protocol HZ-CA-301 (NCT00450658)or Horizon Protocol HZ-CA-303 (NCT00450216)
Brief Title: Double-Blind Follow-on Safety Study of HZT-501 (Ibuprofen 800 mg/Famotidine 26.6 mg) in Subjects Who Have Completed Participation in HZ-CA-301 (NCT00450658) or HZ-CA-303 (NCT00450216)
Acronym: HZ-CA-304
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HZ-CA-304
Record Dates: First submitted 2008-01-28; First posted 2008-02-12 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Chronic Low Back Pain; Chronic Regional Pain Syndrome; Chronic Soft Tissue Pain
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Complex Regional Pain Syndromes | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HZT-501 (Experimental): HZT-501: ibuprofen 800mg/famotidine 26.6mg
  Interventions: Drug: HZT-501
- Ibuprofen (Active Comparator): Ibuprofen 800mg
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: HZT-501 — Ibuprofen 800mg/famotidine 26.6 mg administered orally 3 times daily for 2 weeks
  Arms: HZT-501
Drug: Ibuprofen — Ibuprofen 800mg administered orally 3 times daily for at least 28 weeks
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to evaluate the safety of long-term treatment with HZT-501.

DETAILED DESCRIPTION:
Subject who have completed the 24-week Treatment Period of Horizon Protocol HZ-CA-301 or HZ-CA-303 without developing an upper gastrointestinal ulcer and who are expected to continue to require daily administration of an NSAID for the next 6 months will receive treatment with the same study medication received while participating in HZ-CA-301 or HZ-CA-303.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Expected to continue to require daily administration of an NSAID for at least the coming 6 months.
* Subject completed the 24-week Treatment period of either Horizon Protocol HZ-CA-301 or HZ-CA-303

Exclusion Criteria:

* Subject didn't meet all of the Inclusion and Exclusion Criteria for Horizon Protocol HZ-CA-301 or HZ-CA-303
* Subject developed or experienced any of the following while on either HZ-CA-301 or HZ-CA-303
* Malignant Disease of the gastrointestinal tract
* Erosive esophagitis
* Clinically significant cardiac, renal or hepatic disease
* Uncontrolled diabetes
* Positive pregnancy test on Study Day 0
* Please note that there are other additional criteria. The study center will determine if you meet all of the criteria.

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- PRA International, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants that completed the 24-week Treatment Period of Horizon Protocol HZ-CA-301 (NCT00450658) or Horizon Protocol HZ-CA-303 (NCT00460216) without developing an upper gastrointestinal ulcer and who were expected to continue to require daily administration of an NSAID for at least the coming six months were eligible to enroll.
Pre-assignment Details: Participants continued to receive treatment with the same double-blind study drug (either HZT 501 [ibuprofen 800 mg/famotidine 26.6 mg] or ibuprofen 800 mg administered TID) they received while participating in Protocol HZ-CA-301 (NCT00450658) or Protocol HZ-CA-303 (NCT00460216).
Groups:
- HZT-501 (Ibuprofen/Famotidine): HZT-501: ibuprofen 800mg/famotidine 26.6mg
Period: Overall Study
Arm/Group | HZT-501 (Ibuprofen/Famotidine) | Ibuprofen
Started | 132 | 47
Completed | 112 | 38
Not Completed | 20 | 9
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 7 | 2
Not completed — misc | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HZT-501 (Ibuprofen/Famotidine) | Ibuprofen | Total
Number analyzed (Participants) | 132 | 47 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 110 | 41 | 151
  >=65 years | 22 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.6) | 53.6 (9.3) | 55.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 32 | 122
  Male | 42 | 15 | 57
Region of Enrollment [Number; unit: participants]
  United States | 132 | 47 | 179

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: The objective of this study was to evaluate the long term safety of HZT-501 (ibuprofen 800 mg/famotidine 26.6 mg). No efficacy analyses were planned or performed. Adverse event information was elicited from each participant by indirect questioning using a non-leading question, such as "Has anything bothered you since your last visit or is anything bothering you now?" Adverse event data may also have been volunteered by the participant to the investigator or designee. Physicians assessed the seriousness, severity and causality of each adverse event.
Time Frame: 28 weeks
Measure: Number; unit: participants
Arm/Group | HZT-501 (Ibuprofen/Famotidine) | Ibuprofen
Number analyzed (Participants) | 132 | 47
participants | 55 | 16
Statistical Analysis 1: Comparison: HZT-501 (Ibuprofen/Famotidine) vs Ibuprofen; Test type: Superiority or Other; p = 0.4228, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: End of Study visit occurred at Week 28. Subjects were contacted by telephone four weeks after administration of their final dose of study drug for follow-up of any AEs and to determine if they had experienced any SAEs.
Arm/Group | HZT-501 (Ibuprofen/Famotidine) | Ibuprofen
Serious Adverse Events (participants affected / at risk) | 3/132 | 2/47
Other Adverse Events (participants affected / at risk) | 55/132 | 16/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HZT-501 (Ibuprofen/Famotidine) (N=132) | Ibuprofen (N=47)
diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
esophageal stenosis (Gastrointestinal disorders) | 0 | 1
non-cardiac chest pain (General disorders) | 1 | 0
cholecystitis (Hepatobiliary disorders) | 1 | 0
cellulitis (Infections and infestations) | 1 | 0
gastroenteritis viral (Gastrointestinal disorders) | 0 | 1
diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1
hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HZT-501 (Ibuprofen/Famotidine) (N=132) | Ibuprofen (N=47)
anemia (Blood and lymphatic system disorders) | 2 | 0
cataract (Eye disorders) | 0 | 1
abdominal pain upper (Gastrointestinal disorders) | 2 | 0
abdominal tenderness (Gastrointestinal disorders) | 0 | 1
constipation (Gastrointestinal disorders) | 2 | 0
diarrhea (Gastrointestinal disorders) | 0 | 1
dyspepsia (Gastrointestinal disorders) | 3 | 0
esophageal stenosis (Gastrointestinal disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 2 | 0
vomiting (Gastrointestinal disorders) | 0 | 1
edema peripheral (General disorders) | 0 | 2
gait disturbance (General disorders) | 0 | 1
non-cardiac chest pain (General disorders) | 1 | 1
cholelithiasis (Hepatobiliary disorders) | 0 | 1
bronchitis (Infections and infestations) | 2 | 1
bronchitis acute (Infections and infestations) | 0 | 1
ear infection (Infections and infestations) | 1 | 1
gastroenteritis viral (Infections and infestations) | 4 | 2
influenza (Infections and infestations) | 4 | 1
laryngitis (Infections and infestations) | 0 | 1
otitis media (Infections and infestations) | 2 | 0
sinusitis (Infections and infestations) | 5 | 0
upper respiratory tract infection (Infections and infestations) | 3 | 1
urinary tract infection (Infections and infestations) | 3 | 0
viral upper respiratory tract infection (Infections and infestations) | 3 | 1
animal bite (Injury, poisoning and procedural complications) | 2 | 0
contusion (Injury, poisoning and procedural complications) | 0 | 1
fall (Injury, poisoning and procedural complications) | 0 | 1
rib fracture (Injury, poisoning and procedural complications) | 0 | 1
diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
diabetes mellitus non-insulin dependent (Endocrine disorders) | 0 | 1
hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 1
hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
hyperlipidemia (Metabolism and nutrition disorders) | 0 | 1
hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
carpal tunnel syndrome (Nervous system disorders) | 2 | 0
dizziness (Nervous system disorders) | 2 | 1
nerve compression (Nervous system disorders) | 0 | 1
anxiety (Psychiatric disorders) | 0 | 1
throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
swelling face (Skin and subcutaneous tissue disorders) | 2 | 0
hypertension (Vascular disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI reserves the right to publish or otherwise make public the Study results provided that such communication occurs only after (i) the results of the multicenter Study in its entirety have been publicly disclosed by, or with consent of the sponsor or (ii) 18 months after conclusion of the Study at all sites, whichever comes first. Following this, PI can publish, present or use any non-confidential study results following Sponsor review. PI will not make public raw data or Case Reports.